CLINICAL TRIAL: NCT01699802
Title: Influence of Inhaled Anaesthetics on Rebreathing of Carbon Dioxide When Using an Anaesthesia Gas Reflector (AnaConDa)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/148
Record Dates: First submitted 2012-09-25; First posted 2012-10-04 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhaled anaesthetic agent (Experimental): The group where the investigators adds inhaled anaesthetic agent when using the anaesthetic gas reflector (AnaConda).
  Interventions: Other: Inhaled anaesthetic agent

INTERVENTIONS:
Other: Inhaled anaesthetic agent

SUMMARY:
The purpose is to investigate how the adsorptive capacity of the active carbon filter to carbon dioxide in an anaesthetic gas reflector (AnaConDa) is affected by adding inhaled anaesthetic agent.

The hypothesis is that addition of inhaled anaesthetic agent will affect the amount of adsorption of carbon dioxide to the active carbon and thereby affect rebreathing of carbon dioxide.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary artery by-pass graft surgery
* elective valve replacement surgery
* normal left ventricular ejection fraction on preoperative echocardiography

Exclusion Criteria:

* obstructive lung disease
* restrictive lung disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Volume of carbon dioxide rebreathing from an anesthetic gas reflector | 2 hours
  Tidal carbon dioxide volume rebreathed from an anesthetic gas reflector correlated to concentration of delivered anesthetic gas.

SECONDARY OUTCOMES:
Quantification of ventilatory requirements to maintain isocapnia with the use of an anesthetic gas reflector. | 2 hours
  Changes of tidal volume required to maintain constant alveolar ventilation will be assessed by continuous measurement of exhaled tidal carbon dioxide volume, the latter to be maintained at a constant value.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Bodelsson, Professor, Principal Investigator — Divison of Surgery, Department of Anaesthesia, Skane University Hospital, Lund, Sweden
Locations (1):
- Skane University Hospital Lund, Cardiothoracic Intensive Care, Lund, Sweden